CLINICAL TRIAL: NCT03349762
Title: A Real-World Study Investigating Huaier Granules for Prevention of Recurrence and Metastasis of Colorectal Cancer Patients Following Radical Surgery
Brief Title: Huaier Granules for Prevention of Recurrence and Metastasis of Colorectal Cancer Patients Following Radical Surgery
Status: Recruiting | Type: Observational
Sponsor: Xi Shan Wang (Other)
Responsible Party: Sponsor-Investigator, Xi Shan Wang, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Other Study IDs: HE-201709
Record Dates: First submitted 2017-11-14; First posted 2017-11-22 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Colorectal Cancer
Keywords: Huaier Granule; multisite; open-label; prospective
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Observational 1: Radiotherapy or Chemotherapy
- Observational 2: Huaier Granule & Radiotherapy or chemotherapy
- Observational 3: Huaier Granules

SUMMARY:
To evaluate the efficacy and safety of Huaier granules for Prevention of Recurrence and Metastasis of colorectal cancer patients following radical surgery

DETAILED DESCRIPTION:
This is a multisite, open-label, prospective study investigating Huaier Granule for Prevention of Recurrence and Metastasis of colorectal cancer patients following radical surgery，to evaluate the efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ages 18-75 years;
2. The first time to the therapy of patients who received the radical surgery within two months, Postoperative histopathology confirms the diagnosis of colorectal cancer with stage IIB, IIC and III ( TNM classification)
3. ECOG score of 0-2;
4. No history of malignant tumors;
5. The patients are volunteered for the study, sign informed consent form and cooperate with Investigator to collect data.

Exclusion Criteria:

1. Patients have basic diseases including heart diseases, cerebrovascular disease, lung disease, severe hypertension or diabetes with poor glycemic control;
2. confirmed infections after surgery ;
3. Patients who have post-surgery complications or who are currently under the influence of the radical surgery for colorectal cancer;
4. Being infected with syphilis or with other blood-borne infectious diseases;
5. Pregnancy or lactation; or women of childbearing potential not using contraception;
6. Patients who have taken Traditional Chinese Medicines with efficacy and indications similar to that of Huaier granule - including, but not limited to, compound Banmao capsule., Huachansu capsule, Kangai Injection and Pingxiao tablets;
7. Patients who are suffering from mental illness or Conditions that are considered not suitable for this study investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer patients after radical surgery
Sampling Method: Non-Probability Sample
Enrollment: 3060 (Estimated)
Dates: Start 2018-11-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival(DFS) | 36 months
  Disease free survival (DFS) was defined as the time from participation to the time of tumor recurrence or death.
Overall survival(OS) | 36 months
  OS was defined as the time from participation to death from any cause or last patient last visit.
Local recurrence-Free Survival rate | 36 months
  The proportion of Local recurrence-Free Survival subjects to the total number of subjects.
Distant Metastasis-Free Survival rate | 36 months
  The proportion of Distant Metastasis-Free Surviva subjects to the total number of subjects.

SECONDARY OUTCOMES:
Change From Baseline in Quality of Life (QOL) | 36 months
  Quality of Life (QOL) were measured using supplemental quality of life questions. Item score range（12 items）: 1 (worst symptom) to 5 (no symptom). Change: score at 36 months minus score at baseline.
Incidence rate of Adverse events (AE) | 36 months
  An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Severity of Adverse events | 36 months
  An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Immunity function | 36 months
  Immunity function was measured with Immune cells counts and positive rate.

CONTACTS AND LOCATIONS:
Overall Officials: Xishan Wang, Professor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (22):
- China (22):
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Clinical Hospital affiliated to Harbin Medical University, Harbin, Heilongjiang
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Hubei Cancer Hospita, Wuhan, Hubei
  - Union Hospital Tongji College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Anshan Cancer Hospital, Anshan, Liaoning
  - Ansteel Group General Hospital, Anshan, Liaoning
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - Shandong Provincial Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Zaozhuang Municipal Hospital, Zaozhuang, Shandong
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Fudan University Shanghai Cancer Center, Shanghai